CLINICAL TRIAL: NCT05952752
Title: Effect of Dexamethasone Versus Dexmedetomidine on Postoperative Shivering After Cesarean Section Under Spinal Anesthesia
Brief Title: Dexemedetomidine on Shivering Cesarean Section Under Spinal Anesthesia A Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ayman Abd El-Khalek Mohammed Glala, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: dexemedetomidine on shivering
Record Dates: First submitted 2023-07-02; First posted 2023-07-19 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Postoperative Shivering
Keywords: Dexmedetomidine; Dexamethasone; Postoperative shivering; Shivering; Postoperative analgesia; PONV
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Dexamethasone

STUDY DESIGN:
Intervention Model Description: The estimated sample size for each group was 164 patients. We added 10 % of patients as expected dropout rate. So, the final sample size will be 191 patients per group. Sample size was calculated using G Power 3.1.6.9 (Kiel University, Germany).
  The present study will include American Society of Anesthesiology (ASA) I-II women scheduled for elective CS under intrathecal anesthesia. All patients will be instructed, prepared and monitored according the standard guidelines.
  Preoperative medications will include IV granisetron 1gm and ranitidine 50mg. Spinal anesthesia will be accomplished using 10-12 mg of 0.5% hyperbaric bupivacaine. When adequate level of anesthesia is guaranteed, CS is started under appropriate hemodynamic monitoring. Once the baby is delivered, 10 IV units of oxytocin will be administered. Patients in the studied groups will receive either or intravenous DEXM 10 µg (Sween et al., 2021) or IV infusion of DEXA 8 mg (Esmat et al., 2021).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients in each study category will be equally and randomly assigned to receive either DEXA or DEXM using computer generated random tables and sealed envelopes. Independent researchers who aren't aware of the scope of the study will be assigned to assess and report patient outcome. Used medications will be prepared in similar packages to secure adequate blinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexamethsone (Placebo Comparator): 4 mg will be given for this group IV
  Interventions: Other: Dexamethsone IV
- Dexemedetomidine (Experimental): 12 ug will be given IV infusion for this group
  Interventions: Other: giving dexemedetomidine 12 microgram Iv dripping

INTERVENTIONS:
Other: giving dexemedetomidine 12 microgram Iv dripping — Patients in the studied groups will receive either or intravenous Dexemedetomidine 12 µg
  Other Names: Dexemedetomidine
  Arms: Dexemedetomidine
Other: Dexamethsone IV — 4 mg IV dexamethasone
  Other Names: Dexamethasone
  Arms: Dexamethsone

SUMMARY:
Participants will examine dexemedetomidine versus dexamethasone on postoperative shivering after spinal anesthesia for caesarean section

DETAILED DESCRIPTION:
Patients and Methods Setting and ethics and trial registration The present randomized clinical study is planned to be conducted at Gynecology and Obstetrics Department, Assiut University Hospitals in the time from February through March, 2023. The study protocol will be approved by the independent institutional review board and all participants with provide informed consent prior to enrollment. The study will be registered at clinicaltrials.gov before recruitment of the first patient. Sample size calculation To detect a 20 % of differences between shivering scores in the studies groups, the sample size was calculated using a study power of 95.0 % and two-sided significance level of 5.0 % with 1:1 ratio. The estimated sample size for each group was 164 patients. We added 10 % of patients as expected dropout rate. So, the final sample size will be 191 patients per group. Sample size was calculated using G Power 3.1.6.9 (Kiel University, Germany).

Patient recruitment The present study will include American Society of Anesthesiology (ASA) I-II women scheduled for elective CS under intrathecal anesthesia. Patients will be excluded if they had local infection, bleeding disorder or known allergy to any of the study medications.

Randomization, blinding and allocation Patients in each study category will be equally and randomly assigned to receive either DEXA or DEXM using computer generated random tables and sealed envelopes. Independent researchers who aren't aware of the scope of the study will be assigned to assess and report patient outcome. Used medications will be prepared in similar packages to secure adequate blinding.

Preoperative preparation, monitoring and anesthesia All patients will be instructed, prepared and monitored according the standard guidelines.

Preoperative medications will include IV granisetron 1gm and ranitidine 50mg. Spinal anesthesia will be accomplished using 10-12 mg of 0.5% hyperbaric bupivacaine. When adequate level of anesthesia is guaranteed, CS is started under appropriate hemodynamic monitoring. Once the baby is delivered, 10 IV units of oxytocin will be administered.

Study interventions Patients in the studied groups will receive either or intravenous DEXM 10 µg (Sween et al., 2021) or IV infusion of DEXA 8 mg (Esmat et al., 2021). Outcome assessment The primary outcome of the present study is the incidence of clinically significant postoperative shivering (Grade 2/3) assessed by 4-point scale (Badjatia et al., 2008) as follows:

1. None (Grade 0): no shivering noted on palpation of the masseter, neck, or chest wall
2. Mild (Grade 1): shivering localized to the neck and/ or thorax only
3. Moderate (Grade 2): shivering involved gross movement of the upper extremities (in addition to neck and thorax)
4. Severe (Grade 3): shivering involved gross movements of the trunk and upper and lower extremities Secondary outcome measures will be postoperative pain, hypotension, sedation grade, patient satisfaction, time to sensory and motor onset and time to use of first rescue analgesia.

Statistical analysis All reported data will be recorded and statistically analyzed using appropriate statistical tests.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Pregnant full term
* Undergoing Cesarean section
* Spinal anesthesia

Exclusion Criteria:

* Patient refusal
* General anesthesia
* Contraindications for spinal anesthesia
* Obstetric hemorrhagic complications as placenta accreta, previa, concealed hemorrhage
* Hysterectomy

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 382 (Actual)
Dates: Start 2023-07-20 (Actual); Primary Completion 2023-09-25 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Prevention of postoperative shivering according to bedside shivering assessment scale | till end of spinal anesthesia up to 6 hours
  * grade I: no shivering (score 0)
  * Grade II: localized to the neck or thorax mainly (score 1)
  * Grade III: moderate shivering including the gross length of upper extremeties(score2)
  * Grade IV:severe shivering including the gross movement of the trunk, upper and lower extremities( score 3)

SECONDARY OUTCOMES:
postoperative analgesia according to numerical rating scale( NRS) | 6 hours after induction of spinal anesthesia
  NRS score assessment in combination to time to first rescue of analgesia including score 1 with the least pain experienced in life and score 10 as the most painful experienced pain in life then the pain grading is in between

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university faculty of medicine, Asyut, Asyut Governorate, Egypt